CLINICAL TRIAL: NCT07121010
Title: Randomized Crossover Trial of Protein Source and Leucine Supplementation on Metabolic and Immune Signaling Pathways
Brief Title: How Animal and Plant Protein Shakes Change the Body's Nutrient and Health Responses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ali Ajam, Postdoctoral Associate, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25060010
Record Dates: First submitted 2025-07-16; First posted 2025-08-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Cardiometabolic Health
Keywords: mTOR Signaling; Dietary Protein; Cardiometabolic Disease; Atherosclerosis; Nutrient Signaling
MeSH Terms: conditions — Atherosclerosis | interventions — Leucine

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover study in which each participant receives all three interventions (animal protein smoothie, plant protein smoothie, plant protein smoothie with leucine) on separate study visits in a randomized order. This design allows within-subject comparisons of postprandial responses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal → Plant → Plant+Leucine (Experimental): Participants in this arm will receive the animal-based protein smoothie during their first visit, the plant-based protein smoothie during their second visit, and the plant-based protein smoothie with added leucine during their third visit. All study visits follow the same protocol, including fasting, blood draws, and postprandial assessments.
  Interventions: Dietary Supplement: Animal-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie with Leucine
- Plant-Based → Plant-Based with Leucine → Animal-Based (Experimental): Participants in this arm will receive the plant-based protein smoothie first, the plant-based protein smoothie with leucine second, and the animal-based protein smoothie third. All clinical procedures are the same across visits.
  Interventions: Dietary Supplement: Animal-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie with Leucine
- Plant-Based with Leucine → Animal-Based → Plant-Based (Experimental): Participants in this arm will receive the plant-based protein smoothie with leucine at their first visit, the animal-based smoothie second, and the plant-based protein smoothie third. The same procedures will be followed at each visit.
  Interventions: Dietary Supplement: Animal-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie; Dietary Supplement: Plant-Based Protein Smoothie with Leucine

INTERVENTIONS:
Dietary Supplement: Animal-Based Protein Smoothie — This smoothie is formulated to deliver 50% of its total caloric content from high-quality animal-based protein, such as whey protein isolate or pasteurized egg whites. It is designed to evaluate the postprandial metabolic and immune response to animal-derived protein sources. The smoothie does not contain any added free amino acids and is prepared in a food-safe certified kitchen under standardized conditions. All participants consume the smoothie after an overnight fast to ensure consistency in metabolic assessment.
Dietary Supplement: Plant-Based Protein Smoothie — This smoothie is formulated to deliver 50% of its total caloric content from plant-based protein, such as pea or rice protein isolate. It is designed to evaluate the postprandial metabolic and immune response to plant-derived protein sources. The smoothie does not contain any added free amino acids and is prepared in a food-safe certified kitchen under standardized conditions. All participants consume the smoothie after an overnight fast to ensure consistency in metabolic assessment.
Dietary Supplement: Plant-Based Protein Smoothie with Leucine — This smoothie is formulated to deliver 50% of its total caloric content from plant-based protein, using sources such as pea or rice protein isolate. In addition, it is supplemented with pharmaceutical-grade leucine to match the leucine content typically found in animal-based protein sources. The smoothie is designed to assess whether leucine supplementation can modulate the postprandial metabolic and immune response to plant-derived protein. It is prepared in a food-safe certified kitchen and consumed after an overnight fast to maintain consistency across study conditions.

SUMMARY:
The goal of this clinical trial is to learn how different protein types affect the body's metabolism and immune system in healthy adults. The main questions it aims to answer are:

Does drinking smoothies with animal-based or plant-based protein change the level of amino acids like leucine in the blood?

Does adding leucine to a plant-based smoothie make the body respond like it does to an animal-based smoothie?

Participants will:

Come to the research clinic for 3 study visits

Drink a high-protein smoothie at each visit (one with animal protein, one with plant protein, and one with plant protein + leucine)

Give blood samples before and 1 and 3 hours after each smoothie

Researchers will look at how the body's metabolism and immune system respond. They are especially interested in a pathway called mTOR, which helps control how cells use nutrients and may be involved in heart disease like atherosclerosis.

All smoothies are prepared to meet Halal and Kosher dietary guidelines.

DETAILED DESCRIPTION:
This is a randomized, controlled, crossover clinical trial designed to investigate the acute effects of dietary protein source and leucine supplementation on circulating amino acids and downstream metabolic and immune signaling pathways in healthy adults. The study is being conducted by researchers at the University of Pittsburgh and is based on emerging evidence that dietary protein composition-particularly the type and amount of amino acids such as leucine-may influence key biological processes associated with cardiometabolic health.

Proteins are an essential part of the human diet, and different protein sources (plant vs. animal) contain varying amounts and types of amino acids. One amino acid of particular interest is leucine, a branched-chain amino acid (BCAA) known to activate the mTOR (mechanistic target of rapamycin) signaling pathway. The mTOR pathway plays a critical role in regulating cell growth, metabolism, immune responses, and energy use. Excessive or chronic activation of this pathway has been implicated in cardiometabolic diseases, including atherosclerosis, obesity, insulin resistance, and inflammation.

Animal-derived proteins such as milk or meat tend to be richer in leucine than plant-derived proteins like soy or pea protein. This difference may explain some of the metabolic disparities observed between diets high in animal protein versus plant protein. While plant-based diets are often recommended for their anti-inflammatory and cardiovascular benefits, they may lack sufficient leucine to activate anabolic signaling pathways in certain tissues. It remains unclear whether supplementing plant-based protein with free leucine can achieve the same biological responses as animal protein ingestion.

The trial includes three study arms: (1) a smoothie containing only plant-based protein, (2) a smoothie containing animal-based protein, and (3) a plant-based smoothie with added free leucine. Each smoothie is isocaloric and matched in macronutrient content, differing only in protein source and leucine content. All meals will be prepared and administered under controlled conditions at the Clinical and Translational Research Center (CTRC) at UPMC Montefiore.

Participants will be healthy adults without chronic illnesses or recent infections, aged 18 years and older. Each participant will complete all three study visits in a randomized order, with a minimum 3-day washout period between visits. At each visit, participants will be asked to fast for 10 hours overnight before arriving at the CTRC in the morning. Upon arrival, fasting blood will be collected, followed by consumption of the assigned test smoothie. Additional blood samples will be collected at 1 and 3 hours post-consumption to evaluate postprandial responses.

Blood samples will be analyzed for:

Circulating amino acid levels (primary: leucine)

mTORC1 signaling activity in peripheral blood mononuclear cells (PBMCs), assessed via phosphorylation of S6 kinase (pS6)

Inflammatory and immune signaling markers (e.g., IL-6, NF-κB)

Exploratory transcriptomic profiling and broader amino acid analysis if resources allow

The main hypotheses are:

Animal-based protein will induce higher postprandial leucine levels and stronger mTORC1 activation than plant-based protein.

Supplementation of free leucine in the plant-based smoothie will mimic the biological effects of the animal protein smoothie on immune/metabolic responses.

The findings from this study could provide novel insights into how different dietary proteins modulate nutrient sensing and immune pathways. If plant-based protein supplemented with leucine proves to mimic the effects of animal protein, this could support more sustainable and heart-healthy dietary recommendations without compromising key metabolic functions.

Ultimately, this study will contribute to a deeper understanding of the nutritional regulation of mTOR and inflammation in humans and may inform future dietary interventions aimed at preventing or mitigating chronic cardiometabolic diseases such as atherosclerosis and diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. BMI 18.5-29.9 kg/m²
3. Generally healthy, without known chronic illness and/or treatment with chronic medications
4. Willing to comply with dietary restrictions and study procedures
5. Not currently following a prescribed or restrictive diet (for example, vegan, ketogenic or high-protein regimen) or regularly taking high-protein supplements

Exclusion Criteria:

1. History of cardiovascular disease, diabetes, or autoimmune disorders
2. Active use of anti-inflammatory, immunomodulatory, or lipid-lowering medications
3. Renal or hepatic dysfunction
4. Pregnancy or breastfeeding
5. Allergies or intolerances to components of study meals. A list of the smoothie ingredients will be sent to the potential participant with the mailing of the consent form
6. Participation in another interventional study within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Circulating Serum Leucine Concentration | From enrollment to final blood draw at 4 weeks
  This outcome measures the change in circulating serum leucine concentration from fasting baseline to 1 and 3 hours postprandially following ingestion of each of the three test meals: animal-based protein, plant-based protein, and plant-based protein supplemented with free leucine. Values will be compared within participants across the three meal conditions to assess how protein source and leucine content affect postprandial amino acid levels. Serum leucine will be quantified using targeted mass spectrometry.
  Unit of Measure:
  Micromoles per liter (μmol/L)

SECONDARY OUTCOMES:
Change in Monocyte mTORC1 Signaling Activity | From enrollment to final blood draw at 4 weeks
  This outcome measures the change in mTORC1 signaling activity in peripheral blood mononuclear cells (PBMCs) from fasting to 1 and 3 hours after meal ingestion. mTORC1 activation will be quantified by assessing phosphorylation of S6 kinase (pS6K) using flow cytometry and/or Western blotting. Results will be compared within participants across the three dietary interventions-animal-based protein, plant-based protein, and plant-based protein supplemented with leucine-to determine the effect of protein source and leucine content on monocyte nutrient sensing.
  Unit of Measure: Relative band intensity (Western blot) or % pS6+ cells (flow cytometry)
Change in Serum IL-6 Concentration | From enrollment to final blood draw at 4 weeks
  Serum IL-6 concentration will be measured using ELISA to evaluate the inflammatory response to different protein sources and leucine supplementation.
  Unit of Measure:
  pg/mL
Change in Serum TNF-α Concentration | From enrollment to final blood draw at 4 weeks
  Serum TNF-α concentration will be measured using ELISA to evaluate the inflammatory response to different protein sources and leucine supplementation.
  Unit of Measure:
  pg/ml
Change in Serum C-Reactive Protein (CRP) Concentration | From enrollment to final blood draw at 4 weeks
  Serum CRP concentration will be measured using ELISA to evaluate the inflammatory response to different protein sources and leucine supplementation.
  Unit of Measure:
  mg/L

OTHER OUTCOMES:
Exploratory Change in Additional Serum Amino Acid Concentrations | From enrollment to final blood draw at 4 weeks
  If budget and sample quality allow, additional serum amino acids beyond leucine will be measured using targeted mass spectrometry to evaluate broader metabolic responses to dietary protein source and leucine supplementation.
  Unit of Measure:
  μmol/L
Exploratory Change in PBMC Gene Expression Profiles | From enrollment to final blood draw at 4 weeks
  If resources permit, transcriptomic profiling of peripheral blood mononuclear cells (PBMCs) will be performed to assess dietary protein-induced changes in expression of metabolic and inflammatory gene pathways.
  Unit of Measure:
  log₂ fold change

CONTACTS AND LOCATIONS:
Overall Officials: Babak Razani, MD-PhD, Study Director — University of Pittsburgh
Locations (1):
- UPMC Montefiore - Clinical and Translational Research Center (CTRC), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share individual participant data (IPD) or specimens outside the research team. All data collected during the study will be securely stored and maintained by the University of Pittsburgh research team in compliance with institutional data security standards. De-identified data or biospecimens may be used for future research within the institution or shared with collaborators only under appropriate data use or material transfer agreements and with required regulatory approvals.